CLINICAL TRIAL: NCT00791960
Title: Prophylactic Dimenhydrinate for Intraoperative Nausea and Vomiting: A Randomized, Double Blind, Placebo-Controlled Trial
Brief Title: Prophylactic Dimenhydrinate for Intraoperative Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Dr. Jose C.A. Carvalho, Mount Sinai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-01; 08-0206-A
Record Dates: First submitted 2008-11-13; First posted 2008-11-17 (Estimated); Last update posted 2010-03-29 (Estimated); Status verified 2010-03

CONDITIONS: Nausea; Vomiting
Keywords: Cesarean Section; Dimenhydrinate; Gravol; Antiemetics
MeSH Terms: conditions — Nausea; Vomiting | interventions — Dimenhydrinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dimenhydrinate (Active Comparator): Dimenhydrinate
  Interventions: Drug: Dimenhydrinate
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dimenhydrinate — single dose, 25mg, IV, diluted in 9.5mL normal saline.
  Other Names: Gravol
  Arms: Dimenhydrinate
Other: Placebo — single dose, 10 mL normal saline, IV
  Arms: Placebo

SUMMARY:
The purpose of this study will be to determine whether an intravenous dose of dimenhydrinate (also known as Gravol), given before the induction of spinal anesthesia, will decrease the incidence of intraoperative nausea and vomiting in patients undergoing Cesarean delivery.

This medication is commonly given during and after the surgery if required, but it is not known whether a preventative dose will decrease the overall incidence of these side effects.

DETAILED DESCRIPTION:
Nausea and vomiting remain one of the most common complications of Cesarean delivery. The results of this study will show whether or not we can improve our present anesthesia regimen, and improve the satisfaction of patients undergoing Cesarean deliveries, by reducing the incidence of nausea and vomiting. Our current practice is not to use any medication for preventing nausea and vomiting unless required. However, nausea and vomiting come quite fast and unexpectedly during the operation, and most of the time the medication we give does not work fast enough. We are planning to study the anti-nausea medication dimenhydrinate (commonly known as Gravol), which has been safely and widely used during pregnancy, labour and Cesarean deliveries, hoping that its use will decrease the incidence of this unpleasant occurrence.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing elective Cesarean deliveries under spinal anesthesia.
* All patients who gave written informed consent to participate in this study.
* ASA I and II patients.
* Full term normal pregnancy.

Exclusion Criteria:

* All patients who refuse to give written informed consent.
* All patients who claim allergy or hypersensitivity to dimenhydrinate.
* Patients with history of vomiting within 24 hours prior to Cesarean delivery.
* Patients with history of gastrointestinal or psychiatric diseases and morbid obesity
* Patients receiving any of the following drugs within 24 hours before the study: opioids, antiemetics, H2 antagonists, phenothiazine and corticosteroids.
* Patients with severe pregnancy induced hypertension

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 149 (Actual)
Dates: Start 2008-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Incidence of pre or post-delivery nausea as reported by the patient. Nausea will be defined as a subjectively unpleasant sensation associated with urge to vomit. | 2 hours

SECONDARY OUTCOMES:
Severity of nausea, assessed by visual analog scale (1-10) | 2 hours
Presence or absence of retching or vomiting. | 2 hours
Patient sedation as measured by the Ramsay sedation scale. This will be recorded preoperatively, intraoperatively and postoperatively. | 2 hours
Type and amount of any rescue antiemetic medication used. | 2 hours
Newborn Apgar scores at 1 and 5 minutes, as well as any NICU admission. | 2 hours
Technique of uterine closure (exteriorization vs. in-situ repair). | 30 minutes
Dose of opioid used as supplemental intravenous analgesia. | 2 hours
Number of episodes of hypotension. | 2 hours
Occurence of side effects: tachycardia, dizziness, restlessness, dry mouth, and desaturation. | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Griffiths JD, Gyte GM, Popham PA, Williams K, Paranjothy S, Broughton HK, Brown HC, Thomas J. Interventions for preventing nausea and vomiting in women undergoing regional anaesthesia for caesarean section. Cochrane Database Syst Rev. 2021 May 18;5(5):CD007579. doi: 10.1002/14651858.CD007579.pub3. PMID 34002866